CLINICAL TRIAL: NCT06412952
Title: 68Ga-NOTA-RM26 PET/CT in Glioma Patients
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCH-68Ga-RM26 in Glioma
Record Dates: First submitted 2024-04-26; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma | interventions — 68Ga-NOTA-RM26

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-RM26, PET/CT (Experimental): Inject 68Ga-Pentixafor and then perform PET/CT scan.
  Interventions: Drug: 68Ga-RM26

INTERVENTIONS:
Drug: 68Ga-RM26 — Intravenous injection of one dosage of 74-185 MBq(2-5 mCi) 68Ga-RM26. Tracer doses of 68Ga- RM26 will be used to image lesions of glioma by PET/CT.
  Other Names: 68Ga-GRPR antagonist

SUMMARY:
The aim of this study was to investigate the value of 68Ga-NOTA-RM26, an antagonist targeting gastrin-releasing peptide receptor (GRPR) PET tracer, in the diagnosis of high WHO grade glioma and prediction the grade of glioma using positron-emission tomography/computed tomography (PET/CT).

DETAILED DESCRIPTION:
The gastrin-releasing peptide receptor (GRPR), also known as bombesin receptor subtype II (BB2), is a member of the G protein-coupled receptor family of bombesin receptors. GRPR is over-expressed in various types of human tumors including breast cancer. RM26, a GRPR antagonist with high affinity, was discovered by peptide backbone modification of bombesin analogues.To target gastrin-releasing peptide receptor in neoplastic cells of human breast cancer, peptide NOTA-RM26 was synthesized with a PEG3 linker between NOTA and RM26, and then labeled with 68Ga. An open-label brain PET/ CT study was designed to assess its clinical diagnostic value in patients with glioma.

ELIGIBILITY:
Inclusion Criteria:

* suspected or confirmed untreated glioma patients
* signed written consent.

Exclusion Criteria:

* pregnancy
* breastfeeding
* known allergy against Pentixafor
* any medical condition that in the opinion of the investigator,may
* significantly interfere with study compliance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
SUVmax | through study completion, an average of 1.5 years
  SUVmax of focal lesions are measured on 68Ga-RM26 PET/CT.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Chinese Academy of Medical Science & Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Li Y, Wang R, Chen J, Zhu Z, Wang Y, Ma W. 68Ga-NOTA-RM26 PET/CT in the evaluation of glioma: a pilot prospective study. EJNMMI Res. 2025 Jan 17;15(1):6. doi: 10.1186/s13550-025-01198-7. PMID 39821814
- [Derived] Wang R, Li Y, Li Z, Wang J, Li L, Xiang J, Jia C, Peng X, Wang Y, Ma W, Wang L, Jia W, Chen X, Li D, Zhu Z, Zhang J. Gastrin-Releasing Peptide Receptor Targeting PET/CT With 68 Ga-NOTA-RM26 in the Assessment of Glioma and Combined Multiregional Biopsies. Clin Nucl Med. 2025 Apr 1;50(4):316-323. doi: 10.1097/RLU.0000000000005651. Epub 2025 Jan 14. PMID 39806560